CLINICAL TRIAL: NCT02862132
Title: Predicting Response to Vedolizumab in Pediatric Inflammatory Bowel Diseases (IBD) Including Drug Levels: a Multi-center Prospective Cohort Study, From the Pediatric IBD Porto Group of European Society for Paediatric Gastroenterology, Hepatology and Nutrition (ESPGHAN)
Brief Title: Predicting Response to Vedolizumab in Pediatric Inflammatory Bowel Diseases
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Shaare Zedek Medical Center (Other)
Responsible Party: Principal Investigator, Dr Dan Turner, Head, The Juliet Keidan Institute of Pediatric Gastroenterology, Hepatology and Nutrition, Shaare Zedek Medical Center, Jerusalem, Israel, Shaare Zedek Medical Center
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VEDOKIDS
Record Dates: First submitted 2016-07-31; First posted 2016-08-10 (Estimated); Last update posted 2022-10-25 (Actual); Status verified 2022-10

CONDITIONS: Crohn's Disease; Ulcerative Colitis; Inflammatory Bowel Disease
Keywords: VDZ: Vedolizumab; UC: Ulcerative colitis; CD: Crohn's disease; TDM: Therapeutic drug monitoring
MeSH Terms: conditions — Crohn Disease; Colitis, Ulcerative; Inflammatory Bowel Diseases | interventions — vedolizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Vedolizumab (Experimental): IV Vedolizumab 177mg/m2 Body Surface Area (BSA), max. 300mg Induction regimen: 0,2,6 and then every 8 weeks
  Interventions: Drug: Vedolizumab

INTERVENTIONS:
Drug: Vedolizumab
  Other Names: Entyvio

SUMMARY:
Vedolizumab (VDZ) is a humanized immunoglobulin G1 monoclonal antibody acting against α4β7 integrin which modulates lymphocyte trafficking in the gut.

Results from the adult GEMINI-1 and GEMINI-2 trials demonstrated clinical efficacy in induction and maintenance of remission in both ulcerative colitis (UC) and Crohn's disease (CD), respectively.

Recent real life cohorts in adults support the effectiveness of VDZ in inducing and maintaining remission, both in CD and UC. In pediatrics, there are very limited data on the use of VDZ besides two retrospective case series.

Data on immunogenicity and therapeutic drug monitoring (TDM) of VDZ is conflicting in adults and practically non-existent in children.

The investigators aim to prospectively explore the real life short and longer term outcomes of VDZ in pediatric IBD (including growth) and to develop a prediction model for treatment success based on VDZ trough levels and other clinical and laboratory variables.

DETAILED DESCRIPTION:
This is a multi-center prospective cohort study in which the investigators are aim to enroll 140 children under the age of 18 years, diagnosed with CD, inflammatory bowel disease unclassified (IBDU) or UC (approximately 70 in UC/IBDU and 70 in the CD group) who commenced on Vedolizumab for any reason at the discretion of the treating physician.

Patients will be followed up to 3 years at 8 different time points: week 0, week 2, week 6, week 14, week 30, week 54 (1 year), week 108 (2 years) and week 162 (3 years). Blood work will be collected at each visit during the time of venous access insertion for the drug infusion for serum and stool sample will be collected at visits 0, 14, 30, and 54. In addition, at week 0 and 14 whole blood will be collected into a PaxGene tube for gene expression analysis.

ELIGIBILITY:
Inclusion Criteria:

1. Children under the age of 18 years.
2. IBD Diagnosis
3. Initiating Vedolizumab therapy

Exclusion Criteria:

1. Starting Vedolizumab to prevent post operative recurrence

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 142 (Actual)
Dates: Start 2017-01 (Actual); Primary Completion 2022-01 (Actual); Study Completion 2022-01 (Actual)

PRIMARY OUTCOMES:
Complete remission at week 14 | weeks 14
  As defined by all three criteria:
  i. Steroids and Exclusive enteral nutrition (EEN) (defined as >50% of daily calories with enteral nutrition)- free ii. Clinical remission (i.e. weighted Pediatric Crohn's Disease Activity Index (wPCDAI) <12.5 points in CD, and Paediatric Ulcerative Colitis Activity Index (PUCAI) <10 in UC) iii. CRP lower than 1.5 times upper normal limit (UNL) (may be substituted by Erythocytes Sedimentation Rate (ESR) if CRP missing)
Complete remission at week 30 | weeks 30
  As defined by all three criteria:
  i. Steroids and Exclusive enteral nutrition (EEN) (defined as >50% of daily calories with enteral nutrition)- free ii. Clinical remission (i.e. weighted Pediatric Crohn's Disease Activity Index (wPCDAI) <12.5 points in CD, and Paediatric Ulcerative Colitis Activity Index (PUCAI) <10 in UC) iii. CRP lower than 1.5 times upper normal limit (UNL) (may be substituted by Erythocytes Sedimentation Rate (ESR) if CRP missing)
Complete remission at week 54 | weeks 54
  As defined by all three criteria:
  i. Steroids and Exclusive enteral nutrition (EEN) (defined as >50% of daily calories with enteral nutrition)- free ii. Clinical remission (i.e. weighted Pediatric Crohn's Disease Activity Index (wPCDAI) <12.5 points in CD, and Paediatric Ulcerative Colitis Activity Index (PUCAI) <10 in UC) iii. CRP lower than 1.5 times upper normal limit (UNL) (may be substituted by Erythocytes Sedimentation Rate (ESR) if CRP missing)
Complete remission at week 108 | weeks 108
  As defined by all three criteria:
  i. Steroids and Exclusive enteral nutrition (EEN) (defined as >50% of daily calories with enteral nutrition)- free ii. Clinical remission (i.e. weighted Pediatric Crohn's Disease Activity Index (wPCDAI) <12.5 points in CD, and Paediatric Ulcerative Colitis Activity Index (PUCAI) <10 in UC) iii. CRP lower than 1.5 times upper normal limit (UNL) (may be substituted by Erythocytes Sedimentation Rate (ESR) if CRP missing)
Complete remission at week 162 | weeks 162
  As defined by all three criteria:
  i. Steroids and Exclusive enteral nutrition (EEN) (defined as >50% of daily calories with enteral nutrition)- free ii. Clinical remission (i.e. weighted Pediatric Crohn's Disease Activity Index (wPCDAI) <12.5 points in CD, and Paediatric Ulcerative Colitis Activity Index (PUCAI) <10 in UC) iii. CRP lower than 1.5 times upper normal limit (UNL) (may be substituted by Erythocytes Sedimentation Rate (ESR) if CRP missing)

SECONDARY OUTCOMES:
Steroid and EEN free clinical remission (without the need for normal CRP) using PCDAI or PUCAI score and concomitant medication list. | week 30, week 54, week 108, week 162
Steroid and EEN free clinical response (without the need for normal CRP) using PCDAI or PUCAI score and concomitant medication list. | week 30, week 54, week 108, week 162
Fecal calprotectin levels | week 30, week 54, week 108, week 162
  Levels of calprotectin will be measured in the lab using calprotectin kit.
serum CRP levels | week 30, week 54, week 108, week 162
  CRP levels will be measured in the lab
Rate of loss of response including drug levels | week 30, week 54, week 108, week 162
Steroid dependency (defined as cumulative use of >4 months in a year with at least one need to increase dose while weaning) | week 30, week 54, week 108, week 162
Adverse events | week 30, week 54, week 108, week 162
Measures of mucosal inflammation as available as part of clinical care using endoscopy, imaging or capsule endoscopy. | week 30, week 54, week 108, week 162
Time to induction of remission | week 30, week 54, week 108, week 162
Longitudinal Physician Global Assessment (PGA) | week 30, week 54, week 108, week 162
  PGA will be measured using Visual analogue scale (VAS)
Height velocity as compared with the year prior to commencing VDZ | week 30, week 54, week 108, week 162
Need for surgical interventions (including resections, colectomy, and dilatations) | week 30, week 54, week 108, week 162

CONTACTS AND LOCATIONS:
Overall Officials: Dan Turner, MD, Principal Investigator — Shaare Zedek Medical Center
Locations (15):
- United States (4):
  - Connecticut Children's Medical Center, Hartford, Connecticut
  - Atlantic Children's Health-Goryeb Children's Hospital, Morristown, New Jersey
  - Cohen Children's Medical Center of NY, Northwell, New York, New York
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
- Hvidovre University Hospital, Copenhagen, Denmark
- Our Lady's Children's Hospital Crumlin, Dublin, Ireland
- Israel (7):
  - Rambam Medical Cener, Haifa
  - Wolfson Medical Center, Holon
  - Shaare Zedek Medical Center, Jerusalem
  - Schneider Medical Center, Petah Tikva
  - Sheba Medical Center, Ramat Gan
  - Ichilov, Tel Aviv
  - Assaf Harofeh, Tzrifin
- University Children's Hospital Ljubljana, Ljubljana, Slovenia
- The Royal Hospital for Children Glasgow, Glasgow, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] D'Arcangelo G, Turner D, Ledder O, Orlanski-Meyer E, Broide E, Granot M, Matar M, Hussey S, Yerushalmy-Feler A, Norden C, Miele E, Aloi M. Vedolizumab for extraintestinal manifestations in pediatric inflammatory bowel disease: Results from the VedoKids study. J Pediatr Gastroenterol Nutr. 2026 Feb;82(2):495-502. doi: 10.1002/jpn3.70276. Epub 2025 Nov 18. PMID 41251034
- [Derived] Atia O, Shavit-Brunschwig Z, Lev-Tzion R, Stein R, Broide E, Urlep D, Hyams J, Weiss B, Aloi M, Assa A, Gerasimidis K, Nichols B, Russell RK, Turner D. Maintenance treatment with vedolizumab in paediatric inflammatory bowel disease (VEDOKIDS): 54-week outcomes of a multicentre, prospective, cohort study. Lancet Gastroenterol Hepatol. 2025 Mar;10(3):234-247. doi: 10.1016/S2468-1253(24)00319-4. Epub 2025 Jan 6. PMID 39788134
- [Derived] Atia O, Shavit-Brunschwig Z, Mould DR, Stein R, Matar M, Aloi M, Ledder O, Focht G, Urlep D, Hyams J, Broide E, Weiss B, Levine J, Russell RK, Turner D. Outcomes, dosing, and predictors of vedolizumab treatment in children with inflammatory bowel disease (VEDOKIDS): a prospective, multicentre cohort study. Lancet Gastroenterol Hepatol. 2023 Jan;8(1):31-42. doi: 10.1016/S2468-1253(22)00307-7. Epub 2022 Oct 26. PMID 36306803